CLINICAL TRIAL: NCT03465020
Title: ITALIAN ADULT IMMUNE THROMBOCYTOPENIA (ITP) REGISTRY Investigation on a Dynamic Cohort of Italian Patients With Active ITP
Brief Title: Investigation on a Dynamic Cohort of Italian Patients With Active ITP
Acronym: ITP0918
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Collaborators: Fondazione Progetto Ematologia (Other)
Responsible Party: Sponsor
Other Study IDs: ITP0918
Record Dates: First submitted 2018-03-08; First posted 2018-03-14 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Idiopathic Thrombocytopenic Purpura
Keywords: Idiopathic; Thrombocytopenic; Purpura
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Purpura | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ITP patients: On active treatment
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Safety and efficacy outcomes of patients on different treatments

SUMMARY:
The objective of the study is to produce a dynamic picture of the adult ITP natural history and management in Italy by collecting standardized information retrospective and prospective data of patients in active management through a nation-wide registry.

DETAILED DESCRIPTION:
Primary immune thrombocytopenia (ITP) is an acquired autoimmune disorder affecting both children and adults, characterized by a platelet count below 100 x 109/L in the absence of any underlying disease explaining the thrombocytopenia. Clinical manifestations may be absent or include cutaneous mucosal or organ bleeding, resulting in an overall mortality rate of less than 1-2%.

Previously, 'acute ITP' was used to describe a self-limited form of the disease and 'chronic ITP' to describe the disease if it lasted for more than 6 months. In 2009, a new terminology for ITP was agreed upon based on the duration of the disease. The new terms for ITP are: 'newly diagnosed ITP (from diagnosis to 3 months), 'persistent ITP' (3-12 months) and 'chronic ITP' (lasting for more than 12 months) [2].

Chronic primary ITP in adults is slightly more common in women of childbearing age but the sex incidence is similar in patients over 60. The incidence of ITP in adults is around 4 per 100.000 people per year, with a UK prevalence of up to 24 per 100.000 people [4-6]. No more than 2 per 100.000 will require ITP treatment.

Bleeding is highly variable and there is great heterogeneity. Bleeding is most commonly mucocutaneous, involving the skin and subcutaneous tissue (petechiae, ecchymoses, subcutaneous hematomas), the external mucosae (epistaxis, gum bleeding, blood blisters in the mouth), muscles (muscle hematomata) or the various organs and internal mucosae (hematuria, gastrointestinal bleeding, menorrhagia, intracerebral bleeding). Major bleeding is not common if the platelet count is above 30x109/L. Intracranial hemorrhage is rare and is most often seen in older patients who have additional comorbidities and in patients who fail to respond to therapy. The yearly risk of fatal hemorrhage is around 1.6-3.9% in unresponsive patients. This risk varies with age, from 0.4% per year in patients below 40 years old to 13% per year in those over 60. The natural history of ITP with currently available treatments is not well known. Available data are mostly based on the era when rituximab and thrombopoietin-receptor agonists (TPO-RA) were not in use.

There is a lack reliable data on how recent treatments have modified the course of the disease. Bleeding frequency and severity, complications like infections, thrombosis, ITP-related symptoms like fatigue, etc. are also largely unknown as are women's related issues. Similarly, the cost of treatment for a patient with ITP is not available. Safety and efficacy of specific recent treatments have been measured mostly in industry-sponsored studies. Furthermore, most studies did not conform to the International Working Group (IWG) on ITP recommendations concerning terminology, definitions, outcome criteria and assessment of bleeding.

To the investigator's knowledge, an ITP Registry is ongoing in UK and in Australia and registries are being planned in other European countries with a prospective of creating an international network. The only established international registry, the ITP PARC study, is operative since 2004 but covers different aspects of the disease. The few Italian registries are of regional dimension and are not aligned to collect standardized information in a uniform way.

ELIGIBILITY:
Inclusion Criteria:

* Patients never treated before for whom an ITP treatment is initiated for the first time by the recruiting center
* Patients already treated for whom a new line of ITP treatment is initiated by the recruiting center (the patients could have been treated elsewhere before)
* Patients who, under any ITP treatment at the recruiting center.

Exclusion Criteria:

-Undefined

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All consecutive adult patients (18 years or older) in active treatment for ITP meeting one of the three conditions at their first visit after the enrolment has been opened.
  In all cases, patients should be enrolled at the first visit during the enrolment period (or at latest within 1 month with data referred back to the first visit).
Sampling Method: Probability Sample
Enrollment: 861 (Estimated)
Dates: Start 2018-10-15 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events in ITP adult patients | After 36 months from study enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Rodeghiero, Study Chair — Department of Hematology, S. Bortolo Hospital of Vicenza; Marco Ruggeri, Study Director — Department of Hematology, S. Bortolo Hospital, Vicenza
Locations (26):
- Italy (26):
  - Sc Ematologia E Centro Trapianti Midollo Osseo, Parma, SC
  - Aou Ospedali Riuniti "Umberto I - G.M. Lancisi - G. Salesi"- Ancona - Sod Clinica Ematologica, Ancona
  - Aou Consorziale Policlinico - Bari - Uo Ematologia Con Trapianto, Bari
  - Aou Di Bologna - Policlinico S. Orsola-Malpighi - Uoc Ematologia, Bologna
  - Ao Brotzu, Presidio Ospedaliero A. Businco - Cagliari - Sc Ematologia E Ctmo, Cagliari
  - Ctc U.O Di Ematologia Con Trapianto Di Midollo Osseo - Catania, Capranica
  - Arnas Garibaldi, Po Garibaldi-Nesima - Catania - Uoc Ematologia, Catania
  - Aou Careggi - Firenze - Sod Ematologia, Florence
  - Asst Grande Ospedale Metropolitano Niguarda - Milano - Sc Ematologia, Milan
  - Fondazione Irccs Ca' Granda, Ospedale Maggiore Policlinico - Milano - Ematologia - Padiglione Marcora, Milan
  - Asst Di Monza, Ospedale S. Eugenio - Uo Ematologia E Cta, Monza
  - Ao Di Rilievo Nazionale Antonio Cardarelli - Napoli - Uoc Ematologia Con Trapianto Di Midollo, Napoli
  - Aou Federico Ii - Napoli - Uoc Ematologia, Napoli
  - Aou Maggiore Della Carita' Di Novara - Scdu Ematologia, Novara
  - Aou Policlinico P. Giaccone - Palermo - Uo Ematologia, Palermo
  - Ospedale S.M. della Misericordia - STROKE UNIT, Perugia
  - Asl Di Piacenza, Ospedale "Guglielmo Da Saliceto" - Ematologia E Centro Trapianti, Piacenza
  - Ausl Di Reggio Emilia - Arcispedale Santa Maria Nuova, Irccs - Sc Ematologia, Reggio Emilia
  - Fondazione Policlinico Universitario Agostino Gemelli Irccs - Roma - Area Ematologica, Roma
  - Ente Ecclesiastico Casa Sollievo Della Sofferenza - San Giovanni Rotondo - Ematologia, San Giovanni Rotondo
  - Asl Taranto, Ospedale Ss. Annunziata - Uoc Ematologia, Taranto
  - Aou Città Della Salute E Della Scienza, Ospedale S. Giovanni Battista Molinette - Torino - Sc Ematologia - Università Degli Studi Di Torino, Torino
  - Ente Ecclesiastico Cardinale G. Panico - Tricase - Uo Ematologia, Tricase
  - Azienda Sanitaria Universitaria Integrata Di Trieste - Sc Ematologia, Trieste
  - Asui Di Udine - Presidio Ospedaliero "Santa Maria Della Misericordia" - Clinica Ematologica, Udine
  - Aulss 8 Berica - Ospedale Di Vicenza - Uoc Ematologia, Vicenza

IPD SHARING:
Plan to Share IPD: Undecided